CLINICAL TRIAL: NCT01598883
Title: Understanding "Heparin Resistance" in Cardiac Surgery: Altered Heparin Responsiveness and Its Association With Acute Inflammatory Reactions
Brief Title: Understanding "Heparin Resistance" in Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: rEVO Biologics (Industry)
Responsible Party: Principal Investigator, Greg Koski, Greg Koski, PhD, MD, CPI (Honorary), Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Altered Heparin Responsiveness
Record Dates: First submitted 2012-04-24; First posted 2012-05-15 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Cardiopulmonary Bypass; Altered Heparin Response
MeSH Terms: interventions — Heparin; Antithrombins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT after initial heparin bolus less than 450 (Other): If a patients activated clotting time (ACT) is less than 450 after the bolus dose of heparin (350U/kg) they will be randomized to one of two interventions.
  Interventions: Drug: Heparin; Drug: ATryn
- ACT after first intervention less than 450 (Active Comparator)
  Interventions: Drug: Heparin; Drug: ATryn

INTERVENTIONS:
Drug: Heparin — 150 U/kg
  Other Names: Heparin Sodium
Drug: ATryn — 1000 IU
  Other Names: Antithrombin (recombinant)

SUMMARY:
This study will explore altered heparin responsiveness (AHR) in cardiac surgical patients undergoing cardiopulmonary bypass (CPB) requiring systemic anticoagulation with heparin. The investigators will evaluate the hypothesis that AHR may be directly related to, modulated or mediated by interactions between heparin, antithrombin (AT), the heparin-AT complex, and one or more acute phase proteins. The investigators are particularly interested in identifying patients with "true heparin resistance", that is, patients who demonstrate AHR even after antithrombin-replenishment in the presence of an adequate systemic dose of heparin.

DETAILED DESCRIPTION:
This study uses a prospective, randomized, open-label cross-over design to evaluate the responses to recombinant human AT (rhAT) and/or supplemental heparin for restoration of heparin-responsiveness in the presence of biomarkers of acute inflammation, so called acute phase reactants. Our ultimate goal is, of course, to apply this knowledge to optimize perioperative management of anticoagulation in patients undergoing cardiopulmonary bypass.

We will first identify enrolled patients with altered heparin responsiveness (AHR) as defined by an ACT < 450 seconds (the MGH standard target ACT after the initial dose of heparin for CPB). Patients who achieve an ACT > 450 sec will not enter the randomization phase of the study, their participation in the study will be complete and their routine clinical care will continue unaltered. Those with AHR (post-heparin ACT < 450 sec) will be randomized to receive either supplemental heparin or supplemental AT. Those that fail to achieve an adequate ACT after the first supplementation will cross-over to receive the alternate supplement. Blood samples (totaling at most 20 ml) will be taken at each step to measure heparin level, AT level, AT activity. Once a patient is placed onto cardiopulmonary bypass their participation in the study will be complete.

By design, this study replicates routine clinical management of heparin anticoagulation for cardiopulmonary bypass at the MGH. Most patients (80%) coming to cardiac surgery who will undergo CPB respond adequately to a routine initial bolus dose of heparin (ACT > 450 after 350 U/kg); as noted, subjects in this study that achieve the target ACT will be managed according to routine clinical practice without further testing or intervention.

Under routine care, patients with an inadequate initial response to heparin receive either supplemental heparin (150 U/kg) or pooled human antithrombin (1000 Units), or both. In this study, subjects with inadequate heparin response (ACT < 450) after the initial heparin bolus, will be randomly assigned to two comparison groups; half will receive supplemental heparin (150 U/kg) and half will receive AT (1000 IU). Subjects who fail to respond to their assigned first intervention will cross-over to receive the alternate intervention.

Some subjects may not achieve the target ACT despite receiving both supplemental heparin and AT comprising a group of patients with "true heparin resistance" whose coagulation profiles can be further characterized to better understand the mechanisms of the resistance. These subjects will be considered to have completed the study even though they are not yet on cardiopulmonary bypass and will be managed according to the best clinical judgment of their physicians. They may receive additional heparin, additional AT, fresh-frozen plasma, or any combination of these. These patients may be at risk for thrombotic complications during the post-operative period. Accordingly, when clinically appropriate, these individuals may be referred for further evaluation of their coagulation status, but these evaluations will not be done as part of this study.

This is a pathophysiological risk-factor association study that seeks to better understand the phenomenon of altered heparin responsiveness. Accordingly, there is no specific study endpoint apart from achieving an ACT of > 450 sec. In all enrolled subjects we will measure the levels of three acute phase reactants, Factor VIII, fibrinogen and CRP, heparin levels (anti Xa), AT level (immunofixation) and AT activity after the initial heparin dose. For all subjects who do not achieve and ACT of > 450 we will also measure additional heparin levels (anti Xa), AT level (immunofixation), and AT activity after each intervention in the randomization/crossover phase. The total amount of blood taken for the research-specific laboratory test is less than 20 ml.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac or aortic surgery requiring CPB for which heparin will be used for systemic anticoagulation
* Patients scheduled for urgent surgery who are hemodynamically stable and capable of giving voluntary consent
* Patients with platelet factor 4 antibody positivity (antiPF4+) for whom heparin anticoagulation will be used

Exclusion Criteria:

* Patients for whom heparin will not be used for anticoagulation
* Patients with known congenital AT-deficiency
* Patients with known goat milk allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Altered Heparin Responsivness (AHR) | Participants will be followed from the administration of the initial heparin bolus to being placed on CPB, an average of 15 minutes.
  We will first identify patients with AHR as defined by an ACT <450 seconds (the MGH standard target ACT after the initial dose of heparin for CPB). We will evaluate the hypothesis that AHR may be directly related to, modulated or mediated by interactions between heparin, antithrombin (AT), the heparin-AT complex, and one or more acute phase proteins.

SECONDARY OUTCOMES:
"True Heparin Resistance" | Patients will be followed from the administration of the initial heparin bolus to being placed on CPB, an average of 15 minutes.
  Those with AHR (post-heparin ACT < 450 sec) will be randomized to receive either supplemental heparin or supplemental AT. Those that fail to achieve an adequate ACT after the first supplementation will cross-over to receive the alternate supplement. If patient still fails to achieve an adequate ACT after both supplementations they will be classified as having "True Heparin Resistance".

CONTACTS AND LOCATIONS:
Overall Officials: Greg Koski, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States